CLINICAL TRIAL: NCT03746860
Title: Non-interventional Study on the Safety and Use of Allergy Immunotherapy ACARIZAX® 12 SQ-HDM in Real-life Clinical Practice in Adult Patients With House Dust Mite Allergy in France
Brief Title: N.I.S of AIT in Adult Patients With House Dust Mite Allergy in Real Practice in France
Acronym: CARIOCA
Status: Completed | Type: Observational
Sponsor: ALK-Abelló A/S (Industry)
Collaborators: ITEC Services (Other)
Responsible Party: Sponsor
Other Study IDs: NI-MT-05; ID-RCB:2017-A02668-45 (Other: Comité de Protection des Personnes SUD MEDITERRANNEE IV)
Record Dates: First submitted 2018-11-12; First posted 2018-11-20 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Allergic Rhinitis Due to House Dust Mite; Allergic Asthma Due to Dermatophagoides Farinae; Allergic Asthma Due to Dermatophagoides Pteronyssinus
Keywords: Allergy; Allergic Rhinitis; Allergic Asthma; House Dust Mite; Immunotherapy
MeSH Terms: conditions — Hypersensitivity; Rhinitis, Allergic | interventions — Tablets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Tablet, Dispersible — 1 tablet/day with 12 SQ-HDM per lyo-tablet
  Other Names: ACARIZAX 12 SQ-HDM; Standardised allergen extract from house dust mite

SUMMARY:
Non-interventional study to investigate the safety and tolerability of allergy immunotherapy ACARIZAX® 12 SQ-HDM in real-life clinical practice in adults patients (>18 years) with house dust mite allergy over a period of 12 months.

DETAILED DESCRIPTION:
Condition:

* persistent moderate to severe HDM allergic rhinitis despite use of symptom-relieving medication
* HDM allergic asthma not well controlled by inhaled corticosteroids and associated with mild to severe HDM allergic rhinitis. Patients' asthma status should be carefully evaluated before the initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* At the discretion of the investigator, patient who will be prescribed ACARIZAX® in line with the approved Summary of Product Characteristics (SmPC) and who have been informed, after explicit written explanation and willing to participate in the study by signed consent

Exclusion Criteria:

* Patient who did not have 12 months prior inclusion or have an on-going, House Dust Mite (HDM) Allergy Immunotherapy (AIT).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults suffering of HDM allergic rhinitis or HDM allergic asthma not well controlled by inhaled corticosteroids and associated with mild to severe HDM allergic rhinitis.
  Patients are only included in the study after the decision for treatment with ACARIZAX® has already been made, and only with the objective of documenting data that reflects the treatment and its safety under 'real life' conditions. Accordingly, only examinations and inquiries conforming to routine practice are conducted and documented.
Sampling Method: Non-Probability Sample
Enrollment: 1508 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Safety analysis: Number of patients with at least one Adverse Event | 1 year
  Number of patients with at least one Adverse Events related to ACARIZAX®.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal DEMOLY, Pr, Principal Investigator — Hôpital Arnaud de Villeneuve - 34090 Montpellier - FRANCE
Locations (1):
- Hôpital Arnaud de Villeneuve, Montpellier, France

IPD SHARING:
Plan to Share IPD: No